CLINICAL TRIAL: NCT02667418
Title: CSP #596 - Optimal Treatment for Recurrent Clostridium Difficile Infection
Brief Title: Optimal Treatment for Recurrent Clostridium Difficile
Acronym: OpTION
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study sponsor stopped the trial early after enrolling 308 of the target sample size because of a slower than expected recruitment rate.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 596; #15-03 (Other: VA Central IRB); 1613088 (Other: Hines R&DC)
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Results first posted 2025-11-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Clostridium; Difficile; Fidaxomicin; Vancomycin
Keywords: Clostridium; Difficile; Fidaxomicin; Vancomycin; Recurrent; Pulse; Taper
MeSH Terms: conditions — Recurrence | interventions — Fidaxomicin; Vancomycin; Pulse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Fidaxomicin (Other): Standard 10-day fidaxomicin treatment for Clostridium difficile
  Interventions: Drug: Fidaxomicin
- Vancomycin T/P (Other): Standard 10-day vancomycin treatment followed by taper and pulse vancomycin treatment for Clostridium difficile
  Interventions: Drug: Vancomycin with Taper/Pulse
- Vancomycin (Other): Standard 10-day vancomycin treatment for Clostridium difficile
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Fidaxomicin — 200 mg PO twice daily for 10 days
  Arms: Fidaxomicin
Drug: Vancomycin with Taper/Pulse — 125 mg PO four times daily for 10 days, followed by 125 mg once daily x 7 days, then once every other day x 7 days, then once every 3rd day x 7 days
  Arms: Vancomycin T/P
Drug: Vancomycin — 125 mg PO for times daily for 10 days
  Arms: Vancomycin

SUMMARY:
The purpose of this study is to determine whether fidaxomicin and vancomycin followed by taper and pulse vancomycin treatment are superior to standard vancomycin treatment for the treatment of recurrent Clostridium difficile infection.

DETAILED DESCRIPTION:
Abstract Clostridium difficile is the most common cause of healthcare-associated infectious diarrhea among adults in industrialized countries. In addition to diarrhea, C. difficile infection (CDI) may also result in serious complications such as shock, toxic megacolon, colectomy, and death. The Centers for Disease Control and Prevention (CDC) has estimated C. difficile results in 250,000 hospital infections, 14,000 deaths, and $1 billion in excess costs annually. Recurrent CDI is the most challenging clinical dilemma facing clinicians who treat this disease. An estimated 30% of patients who respond to initial treatment with either vancomycin or metronidazole develop recurrent CDI, usually within 1-4 weeks of completing treatment.

The primary objective of this study is to determine whether 1) standard fidaxomicin treatment and 2) standard vancomycin treatment followed by taper and pulse vancomycin treatment are superior to standard vancomycin treatment alone for sustained clinical response at day 59 for all treatments, for participants with either their first or second recurrence of CDI. Veterans presenting with a first or second CDI recurrence will be screened, consented and randomly assigned in a double-blind manner equally to one of three treatment groups: 1) a 10 day course of oral vancomycin (VAN-TX), 2) a 10 day course of fidaxomicin (FID-TX) or 3) a 31 day course of vancomycin which includes a taper and pulse following daily treatment (VAN-TP/P). Symptom resolution is defined as an improvement or resolution of diarrhea ( 3 unformed bowel movements over 24 hours) for 48 consecutive hours compared to the participant's baseline. Recurrence is defined as having diarrhea (>3 loose or semi-formed stools over 24 hours for 48 consecutive hours). A sample size of 459 randomized study participants is required to obtain 91% global power to detect a 16% absolute difference (expected proportion of 31% in the VAN-TX group) in sustained clinical response (D- COM) proportion for at least one comparison (VAN-TP/P vs. VAN-TX, FID-TX vs. VAN-TX) at the family wised error rate (FWER) 0.05 level. The marginal probability (disjunctive power) of detecting 16% absolute difference for each comparison is 81%. The expected withdrawal rate prior to day 59 (prior outcome assessment) is estimated to be 10%. If both FID-TX and VAN-TP/P are found to be superior to VAN-TX, then the non-inferiority of VAN-TP/P to FID-TX will be assessed.

With the assumption that sites recruit 4 participants (site average) per year for sites primarily recruiting from the main hospital and nearby CBOCS, and 6 participants (site average) per year for sites that could partner with independent VAMCs (Independent VAMCs LSI Application will be reviewed and approved by Central IRB) that are close in distance to allow a shared site coordinator (WOC appointed) at an increased funding level, the study is expected to complete enrollment of 459 participants within 6 years with 90 days of follow-up. This includes 2 years of pilot phase plus transitioning period from pilot phase to full study, and 4 years of full study. There were 6 sites in the pilot phase and will have 24 units (26 sites) in full phase (including 5 pilot sites and 21 additional sites). Sites that are significantly below the recruitment target for an extensive period may be considered for termination. The recruitment timeline and the number of sites will be re-evaluated based on the actual recruitment rate, the number of sites still recruiting, whether replacement or additional sites will be added, the study time period on administrative recruitment hold due to COVID-19 pandemic, and available funding resources.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained and signed
* Age > 18
* If female, participant must not be pregnant or nursing

  * Negative pregnancy test required for females <61 years of age or without prior hysterectomy
* Confirmed current diagnosis of CDI, determined by having

  * >3 loose or semi-formed stools for participants over 24 hours AND
  * Positive stool assay for C. difficile
  * EIA positive for toxin A/B; or
  * Cytotoxin assay; or
  * Nucleic Acid Amplification Test (NAAT, PCR or LAMP) based detection of toxigenic C. difficile
* Current episode represents the first recurrent episode of CDI within 3 months of the primary CDI episode in a patient who has not had CDI in the 3 months prior to the primary episode OR a second recurrent CDI episode occurring within 3 months of the first recurrent episode, as defined above

  * At least one of the previous CDI episodes must have been confirmed by a stool assay for C. difficile

Exclusion Criteria:

* Inability to provide informed consent
* Inability to take oral capsules
* Receipt of >72 hours of antibiotics considered effective in the treatment of CDI, including:

  * metronidazole
  * vancomycin
  * fidaxomicin
  * nitazoxanide
  * rifaximin
* Prior infusion of bezlotoxumab within the previous 6 months
* Known presence of fulminant CDI, including hypotension, severe ileus or GI obstruction or incipient toxic megacolon
* Receipt of more than a single course of oral vancomycin, fidaxomicin, or a vancomycin tapering regimen since the primary episode of CDI as defined above
* Known allergy to vancomycin or fidaxomicin
* Acute or chronic diarrhea due to inflammatory bowel disease or other cause (e.g., presence of an ileostomy or colostomy) that would confound evaluation of response to CDI treatment
* Anticipation of need for long term systemic antibiotic treatment (beyond 7 days)
* Patients with an active diagnosis of COVID-19 will be excluded from the study, but patients who have recovered (per current CDC guidance on discontinuation of transmission-based precautions) can be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart B. Johnson, MD BA, Study Chair — Edward Hines Jr. VA Hospital, Hines, IL; Dale N Gerding, MD, Study Chair — Edward Hines Jr. VA Hospital, Hines, IL
Locations (32):
- United States (31):
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona
  - Central Arkansas Veterans Healthcare System, Little Rock, AR, Little Rock, Arkansas
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Northern California Health Care System, Mather, CA, Sacramento, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Rehabilitation R&D Service, Baltimore, MD, Baltimore, Maryland
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan
  - Asheville VA Medical Center, Asheville, NC, Asheville, North Carolina
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Oklahoma City VA Medical Center, Oklahoma City, OK, Oklahoma City, Oklahoma
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin
- VA Caribbean Healthcare System, San Juan, PR, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson S, Gerding DN, Li X, Reda DJ, Donskey CJ, Gupta K, Goetz MB, Climo MW, Gordin FM, Ringer R, Johnson N, Johnson M, Calais LA, Goldberg AM, Ge L, Haegerich T. Defining optimal treatment for recurrent Clostridioides difficile infection (OpTION study): A randomized, double-blind comparison of three antibiotic regimens for patients with a first or second recurrence. Contemp Clin Trials. 2022 May;116:106756. doi: 10.1016/j.cct.2022.106756. Epub 2022 Apr 7. PMID 35398532

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fidaxomicin | Vancomycin T/P | Vancomycin
Started | 105 | 102 | 101
Modified Intent-To-Treat | 100 | 99 | 100
Safety Set | 102 | 100 | 100
Completed | 84 | 91 | 94
Not Completed | 21 | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fidaxomicin | Vancomycin T/P | Vancomycin | Total
Number analyzed (Participants) | 105 | 102 | 101 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (12.5) | 67.7 (11.9) | 67.9 (12.0) | 67.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 11 | 29
  Male | 93 | 96 | 90 | 279
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One participant in Fidaxomicin with missing race information
  Participants
    White: number analyzed (Participants) | 104 | 102 | 101 | 307
    White | 86 | 80 | 79 | 245
    African American: number analyzed (Participants) | 104 | 102 | 101 | 307
    African American | 15 | 18 | 19 | 52
    Other: number analyzed (Participants) | 104 | 102 | 101 | 307
    Other | 3 | 4 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Clinical Response as Measured at Study Day 59 for All Treatment Regimens
Description: The Primary outcome will be sustained clinical response as measured at study day 59 for all treatment regimens. Sustained clinical response is a composite outcome that includes symptom resolution during treatment without any of the following (as assessed on day 59):
  1. Diarrhea recurrence
  2. Other non-fatal clinical events including severe abdominal pain, toxic megacolon (where diarrhea ceases but is not a beneficial outcome), and colectomy
  3. Death
Time Frame: Day 59 for all treatment regimens.
Population: mITT Primary Analysis: Missing primary outcome D-COM at Day 59 in the mITT analysis was imputed by an imputation model.
  mITT Sensitivity Analysis 1: Missing primary outcome D-COM at Day 59 was treated as failure.
  mITT Sensitivity Analysis 2: Missing outcomes were excluded as a complete case analysis.
  PP analysis: Participants who 1) failed to respond by day 10 or completed day 59 follow-up and (2) took 80% of their assigned drug according to the pill count (Per-Protocol population).
Measure: Count of Participants; unit: Participants
Arm/Group | Fidaxomicin | Vancomycin T/P | Vancomycin
Number analyzed (Participants) | 100 | 99 | 100
Participants
  mITT Primary Analysis | 44 | 58 | 44
  mITT Sensitivity Analysis 1 | 40 | 56 | 42
  mITT Sensitivity Analysis 2: number analyzed (Participants) | 91 | 95 | 95
  mITT Sensitivity Analysis 2 | 40 | 56 | 42
  PP Analysis: number analyzed (Participants) | 83 | 91 | 93
  PP Analysis | 39 | 55 | 42

2. Secondary Outcome: Sustained Diarrhea Composite Outcome (D-COM) at 28 Days Post End of Therapy
Description: Sustained Diarrhea Composite Outcome (D-COM) at 28 days Post End of Therapy- Secondary Analyses of Primary Outcome. Sustained clinical response without recurrent CDI (CDI-COM) at 28 days post end of therapy for all three treatment regimens. Sustained clinical response was defined using the same criteria as previously stated except that the endpoint will be 28 days after the last dose of treatment drug for each treatment arm (day 38 for vancomycin and fidaxomicin, and day 59 for vancomycin taper/pulse).Sustained clinical response is a composite endpoint defined as symptom resolution during treatment without diarrhea recurrence, mortality or other important clinical outcomes at any time during the follow-up period. Those participants failing to meet the criteria of symptom resolution (diarrhea resolution) by the end of the active treatment (day 10 for all groups), or who experience a recurrence during the follow-up period, will be considered study treatment failures.
Time Frame: 28 Days Post End of Therapy
Population: mITT Complete Case Analysis with missing outcome excluded, number of participants in population would be different in other mITT complete case analysis populations because timeline for data collection and outcome variables were different.
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin T/P | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 95 | 92 | 96
Participants | 56 | 51 | 48

3. Secondary Outcome: Clostridium Difficile Infection Composite Outcome (CDI-COM)
Description: Clostridium difficile Infection Composite Outcome (CDI-COM) at day 59 post randomization. Sustained response in CDI-COM is defined using the same composite endpoint criteria as was used in the D-COM composite outcome but with confirmation of no CDI recurrence by a negative C. difficile stool assay test (i.e., proportion of subjects who achieve symptom resolution by day 10 without recurrent CDI, without non-fatal clinical events, and without death).
Time Frame: Day 59 post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin T/P | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 91 | 83 | 91
Participants | 59 | 43 | 44

4. Secondary Outcome: Symptom Resolution
Description: The percentage of participants who had symptom resolution by Day 10 post randomization
Time Frame: Day 10 since randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin T/P | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 97 | 96 | 98
Participants | 90 | 90 | 92

5. Secondary Outcome: CDI Recurrence
Description: CDI recurrence following initial symptom resolution
Time Frame: Day 90 since randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin T/P | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 79 | 68 | 78
Participants | 26 | 29 | 34

6. Secondary Outcome: Diarrhea Recurrence
Description: Diarrhea recurrence with confirmation of recurrent CDI following initial symptom resolution
Time Frame: Day 90 since randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin T/P | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 85 | 77 | 83
Participants | 35 | 41 | 41

7. Secondary Outcome: C.Diff Health Related Quality of Life (HRQOL)
Description: Change in patient reported C.diff Health Related Quality of Life (HRQOL) from baseline (day 0) to day 10. The HRQOL is measured with patient self-reported 32-item questionnaire. The summary measure, CDiff32-QOL, is the total score that sums over 32 individual items with each item rated on a 5-point Likert scale and then transformed to a 100-point scale with higher score indicating better C.diff Health Related QOL in general. The full scale of the HRQOL: 1-5 on a 5-point Likert scale and 0-100 on the 100-point scale; the minimum: 0 on the 100-point scale and maximum value: 100 on the 100-point scale. The summary measure (32 items) range on the 100-point scale: 0-3200.
Time Frame: Day 10 since randomization
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vancomycin T/P | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 102 | 105 | 101
units on a scale | 451.8 (582.0) | 446.6 (419.1) | 543.8 (535.7)

8. Secondary Outcome: C.Diff Health Related Quality of Life (HRQOL)
Description: Change in patient reported C.diff Health Related Quality of Life (HRQOL) from baseline day 0 to day 59. The HRQOL is measured with patient self-reported 32-item questionnaire. The summary measure, CDiff32-QOL, is the total score that sums over 32 individual items with each item rated on a 5-point Likert scale and then transformed to a 100-point scale with higher score indicating better C.diff Health Related QOL in general. The full scale of the HRQOL: 1-5 on a 5-point Likert scale and 0-100 on the 100-point scale; the minimum: 0 on the 100-point scale and maximum value: 100 on the 100-point scale. The summary measure (32 items) range on the 100-point scale: 0-3200.
Time Frame: day 0- day 59
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vancomycin T/P | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 102 | 105 | 101
units on a scale | 902.7 (682.6) | 818.5 (743.0) | 919.8 (654.3)

9. Secondary Outcome: Sustained Clinical Response (D-COM) BI/NAP1/027 Strain as "Yes"
Description: Sustained clinical response (D-COM) at day 59 for subgroups (infection with the BI/NAP1/027 strain (yes) at study enrollment; etc.). The sliced analysis was used to break down the subgroup factors into different sub-levels and then to explore the differences between treatment group (VAN-TP and FDX) and VAN control group at each level.
Time Frame: Day 59 since randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin T/P | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 18 | 9 | 9
Participants | 8 | 3 | 2

10. Secondary Outcome: Diarrhea Recurrence
Description: Diarrhea recurrence with confirmation of recurrent CDI following initial symptom resolution. Diarrhea recurrence and diarrhea recurrence with confirmation of recurrent CDI following initial symptom resolution. Diarrhea (>3 loose or semi-formed stools over 24 hours) over 48 consecutive hours in participants who achieved initial symptom resolution will be recorded separately from sustained clinical response as will confirmed CDI recurrence.
Time Frame: Day 38 since randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin T/P | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 86 | 80 | 85
Participants | 19 | 30 | 37

11. Secondary Outcome: Diarrhea Recurrence
Description: Diarrhea recurrence with confirmation of recurrent CDI following initial symptom resolution
Time Frame: Day 59 since randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin T/P | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 85 | 78 | 83
Participants | 29 | 39 | 41

12. Secondary Outcome: CDI Recurrence
Description: CDI recurrence following initial symptom resolution
Time Frame: Day 38 since randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin T/P | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 82 | 75 | 80
Participants | 12 | 21 | 28

13. Secondary Outcome: CDI Recurrence
Description: CDI recurrence following initial symptom resolution
Time Frame: Day 59 since randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin T/P | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 79 | 71 | 78
Participants | 21 | 28 | 34

14. Secondary Outcome: Sustained Clinical Response (D-COM) With the BI/NAP1/027 Strain no
Description: Sustained clinical response (D-COM) at day 59 for subgroups (infection with the BI/NAP1/027 strain (no) at study enrollment; etc.). The sliced analysis was used to break down the subgroup factors into different sub-levels and then to explore the differences between therapy group (VAN-TP and FDX) and VAN control group at each level.
Time Frame: Day 59 since randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin T/P | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 55 | 50 | 66
Participants | 34 | 21 | 32

15. Secondary Outcome: Sustained Diarrhea Composite Outcome (D-COM) at 90 Days After Randomization
Description: Sustained Diarrhea Composite Outcome (D-COM) at 90 days after Randomization - Secondary Analyses of Primary Outcome
Time Frame: 90 Days After Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin T/P | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 95 | 91 | 95
Participants | 51 | 36 | 42

ADVERSE EVENTS:
Time Frame: 8 years, 6 months
Arm/Group | Fidaxomicin | Vancomycin T/P | Vancomycin
All-Cause Mortality (participants affected / at risk) | 8/102 | 2/100 | 3/100
Serious Adverse Events (participants affected / at risk) | 34/102 | 30/100 | 27/100
Other Adverse Events (participants affected / at risk) | 7/102 | 15/100 | 12/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fidaxomicin (N=102) | Vancomycin T/P (N=100) | Vancomycin (N=100)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (3) | 1 (1)
Mycardinal infection (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
Upper Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1)
death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Physical deconditioning (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 5 (5) | 6 (6) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Sepsis syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract Infection (Infections and infestations) | 2 (2) | 4 (4) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Cardiac valve vegetation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Renal lymphocele (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkaliemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Alcohol withdrawal (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Chronic Obstructive Pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Homeless (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Alcohol detoxification (Surgical and medical procedures) | 2 (10) | 1 (1) | 1 (1)
Amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Intraocular Lens Implant (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Knee Arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Catheterisation cardiac (Investigations) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fidaxomicin (N=102) | Vancomycin T/P (N=100) | Vancomycin (N=100)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) — Mild
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Moderate
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Mild
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Moderate
Dysepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Mild
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Moderate
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) — Mild
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Severe
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Moderate
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Clostridioide difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Moderate
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Mild
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Mild
Hepatic enzyme increased (Investigations) | 1 (1) | 3 (3) | 1 (1) — Mild
White blood cell count (Investigations) | 0 (0) | 0 (0) | 1 (1) — Mild
White blood cell count (Investigations) | 0 (0) | 1 (1) | 0 (0) — Moderate
Alanine aminotransferase (Investigations) | 1 (1) | 2 (2) | 0 (0) — Mild
Aspartate aminotransferase (Investigations) | 0 (0) | 1 (1) | 0 (0) — Mild
Neutrophil count decrease (Investigations) | 0 (0) | 1 (1) | 0 (0) — Severe
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) — Mild
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) — Mild
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Mild
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Moderate
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Moderate
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) — Mild
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) — Moderate
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Mild
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — Moderate

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-11-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT02667418/Prot_002.pdf
  • Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT02667418/SAP_001.pdf